CLINICAL TRIAL: NCT03690219
Title: Prevalence of Acute Injuries in Amateur and Elite Mountain Bikers
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: MTB
Record Dates: First submitted 2018-09-12; First posted 2018-10-01 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Acute Injury in Mountain Biking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The investigators intented to assess the prevalence of acute injuries in amateur and elite mountain bikers.

DETAILED DESCRIPTION:
In order to assess the prevalence of acute injuries in amateur and elite mountain bikers a questionnaire was created in accordance to existing literature. The questionnaire was translated in several languages by bilingual people familiar with mountain biking. The questionnaire focussed on demographic data, training volume, number of races per year, number of injuries since practising mountain biking, wearing of protective gear items and accident mechanism. The survey was conducted during the Swiss Epic Mountain Bike Event in 2017. All riders were asked to voluntarily participate in the survey.

ELIGIBILITY:
Inclusion Criteria:

* mountain bikers participating in the Swiss Epic Mountain Bike Event in 2017

Exclusion Criteria:

* non-participators, non-mountain bikers in the Swiss Epic Mountain Bike Event in 2017

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators included all mountain bikers participating in the Swiss Epic Mountain Bike Event in 2017, who agreed to attend in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, PhD, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland SUPSI
Locations (1):
- SUPSI, Landquart, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stoop R, Hohenauer E, Vetsch T, Deliens T, Clijsen R. Acute Injuries in Male Elite and Amateur Mountain Bikers: Results of a Survey. J Sports Sci Med. 2019 Jun 1;18(2):207-212. eCollection 2019 Jun. PMID 31191089
- See also: fullversion of publication — https://pmc.ncbi.nlm.nih.gov/articles/PMC6543986/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the 2017 Swiss Epic Mountain Bike Event in Valais, riders completed a retrospective survey on bike-related injuries. 99 returned questionnaires were eligible for injury prevalence analysis. For the detailed analysis, 29 riders without injuries and 14 questionnaires with missing data were removed. Ultimately, 56 participants were included in the final analysis.
Pre-assignment Details: To assess eligibile data, incomplete data sets in terms of gender, age, riding level and injury reporting were excluded. In a next step, due to the low number of female respondents, female participants were excluded to ensure comparability and homogeneity of the data.
Groups:
- Elite Mountain Bikers: A group of mountain bikers, attending the Swiss Epic Mountain Bike Event 2017, self-reported their riding level as semi-professional or professional in a questionnaire.
- Amateur Mountain Bikers: A group of mountain bikers, attending the Swiss Epic Mountain Bike Event 2017, self-reported their riding level as recreational or amateur in a questionnaire.
Period: Overall Study
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
Started | 31 | 68
Completed | 15 | 41
Not Completed | 16 | 27
Not completed — no injuries | 9 | 20
Not completed — missing information | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers | Total
Number analyzed (Participants) | 15 | 41 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.47 (12.12) | 40.7 (7.6) | 39.40 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 41 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 15 | 41 | 56

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Injuries in Amateur and Elite Mountain Bikers
Description: In a retrospective questionnaire participants were asked about the "Number of injuries obtained during mountain biking".
Time Frame: At study enrollment, based on participants' self-reported history of mountain bike injuries
Measure: Mean (Standard Deviation); unit: Number of injuries
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
Number analyzed (Participants) | 15 | 41
Number of injuries | 4.6 (5.5) | 3.5 (4.3)

2. Secondary Outcome: Training and Racing Volume
Description: In a retrospective questionnaire the participants were asked "How many races per year" they ride and whats their "Estimated training hours per week in regard to the season".
  The number of races per year was multiplied by the factor 4 to transform the number of races into training hours. Then, both values were added to get the training volume per year.
Time Frame: At study enrollment, based on participants' retrospective self-report of the number of races per year and estimated training hours per week
Measure: Mean (Standard Deviation); unit: hours per year
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
Number analyzed (Participants) | 15 | 41
hours per year | 743.86 (238.12) | 443.1 (214.13)

3. Secondary Outcome: Years Practising Mountain Biking
Description: In a retrospective questionnaire participants were asked "Since how many years do you participate in mountain biking?".
Time Frame: At study enrollment, based on participants' self-reported history of mountain bike participation
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
Number analyzed (Participants) | 15 | 41
years | 15.73 (6.78) | 15.29 (8.89)

4. Secondary Outcome: Amount of Protective Gear Items
Description: In a retrospective questionnaire participants were asked to tick the protective gear (helment, gloves, eveywear, upper armour, lower armout, other) they are using for mountain biking.
Time Frame: At study enrollment, based on participants' retrospective self-report of protective gear use
Measure: Mean (Standard Deviation); unit: amount of worn protective gear items
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
Number analyzed (Participants) | 15 | 41
amount of worn protective gear items | 3.20 (0.77) | 3.24 (0.73)

5. Secondary Outcome: Injury Rate Per 1000hrs Exposure Time
Description: The injury rate per 1000 hours exposure time was calculated as follows: the hours of exposure time per year were multiplied by the number of years practicing mountain biking to get the total hours at risk. Then, the total amount of injuries ever was divided by the total hours at risk, multiplied by 1000 hours to get the injury rate per 1000 hours of exposure time.
Time Frame: At study enrollment, based on participants' self-reported history of mountain bike participation
Measure: Number; unit: injuries per 1000hrs exposure time
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
Number analyzed (Participants) | 15 | 41
injuries per 1000hrs exposure time | 0.39 | 0.52

ADVERSE EVENTS:
Time Frame: Retrospective; events occurring prior to questionnaire completion
Description: Data was generated through a retrospective questionnaire, participants were not assessed for adverse events.
Arm/Group | Elite Mountain Bikers | Amateur Mountain Bikers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03690219/Prot_SAP_000.pdf